CLINICAL TRIAL: NCT07008118
Title: A Phase 1, Open-Label, Multicenter Study of INCA035784 in Participants With Myeloproliferative Neoplasms
Brief Title: A Study to Evaluate INCA035784 in Participants With Myeloproliferative Neoplasms
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCA035784-101
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Myeloproliferative Neoplasms
Keywords: Myeloproliferative Neoplasms; Myelofibrosis; Essential thrombocythemia; CALR mutation
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1a: Dose escalation (Experimental): INCA035784 will be administered at a protocol defined starting regimen in 28-day cycles as monotherapy to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE[s]). Participants with myeloproliferative neoplasm (MPN) will enroll in this group.
  Interventions: Drug: INCA035784
- Part 1b: Dose expansion (Experimental): INCA035784 will be administered as monotherapy at the RDE(s) identified during Part 1a. Participants with myeloproliferative neoplasm (MPN) will enroll in this group.
  Interventions: Drug: INCA035784

INTERVENTIONS:
Drug: INCA035784 — INCA035784 will be administered at protocol defined dose.

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of INCA035784 in participants with myeloproliferative neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of signing the ICF
* ECOG performance status of 0 to 1 for the dose escalation (Part 1a) and 0 to 2 for the dose expansion (Part 1b)
* Documented CALR exon-9 mutation
* Confirmed diagnosis of MPN according to the 2022 ICC criteria:

  * DIPSS+ intermediate-2/high-risk MF with prior JAKi, <20% blasts, and measurable spleen
  * High-risk ET with platelets >450×10⁹/L
* Resistant, refractory, intolerant, or has lost response to ≥1 prior line of therapy for MF and ≥2 prior lines for ET
* No prior stem cell transplant and none planned within 6 months
* Minimum Laboratory Requirements:

  * Platelet count ≥50 × 10⁹/L
  * Absolute neutrophil count ≥1 × 10⁹/L
  * International normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 × upper limit of normal (ULN), unless receiving vitamin K antagonists
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <2.5 × ULN
  * Total bilirubin <2 × ULN
  * Estimated creatinine clearance >45 or >30 mL/min (depending on study part)

Exclusion Criteria:

* Major bleeding or thrombosis (e.g., stroke, DVT, PE) within the past 3 months
* Active or high-risk HBV, HCV, or HIV infection, or other chronic active infections requiring systemic treatment
* Active invasive cancer within the past 2 years, except certain early-stage or low-risk cancers (e.g., resected skin, cervical, thyroid, or prostate cancer)
* Pregnant or unwilling to avoid pregnancy or fathering a child during the study and for a defined period after the last dose.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-03-14 (Estimated); Study Completion 2029-12-14 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  Dose-limiting toxicity will be defined as the occurrence of any of the toxicities as per protocol.
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to approximately 2 years and 90 days
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug up to 90 days after the last dose of study drug.
Number of participants with TEAEs leading to treatment interruption, discontinuation, or delay | Up to approximately 2 years and 90 days
  Number of participants with TEAEs leading to treatment interruption, discontinuation, or delay.

SECONDARY OUTCOMES:
Number of participants with TEAEs leading to dose modification or discontinuation | Up to approximately 2 years and 90 days
  Number of participants with TEAEs leading to dose modification or discontinuation.
Participants with MF: Response using the revised International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) response criteria for myelofibrosis (MF) | Up to approximately 2 years and 90 days
  Defined as the percentage of participants with Response using the revised IWG-MRT and ELN response criteria.
Participants with essential thrombocythemia (ET): Response using the revised IWG-MRT and ELN response criteria for ET | Up to approximately 2 years and 90 days
  Defined as the percentage of participants with Response using the revised IWG-MRT and ELN response criteria.
Participants with myelodysplastic syndrome (MDS)/MPN: Response using the revised IWG-MRT response criteria for MDS/MPN | Up to approximately 2 years and 90 days
  Defined as the percentage of participants with Response using the revised IWG-MRT response criteria.
Participants with symptomatic anemia: Anemia response | Up to approximately 2 years and 90 days
  Anemia response as defined in the protocol.
Participants with spleen volume (SV) ≥ 450 mL at baseline: Percentage of participants achieving spleen volume reduction of ≥ 35% (SVR35) | Week 12 and Week 24
  Defined as percentage of participants with a protocol defined Spleen Volume Reduction of ≥ 35% (SVR35).
Participants with SV ≥ 450 mL at baseline: Percentage of participants achieving spleen volume reduction of ≥ 25% (SVR25) | Week 12 and Week 24
  Defined as percentage of participants with a protocol defined Spleen Volume Reduction of ≥ 25% (SVR25).
Percentage of participants achieving ≥ 50% reduction from baseline of total symptom score (TSS) | Week 12 and Week 24
  Defined as the percentage of participants achieving ≥ 50% reduction from baseline of TSS.
Mean change from baseline in TSS | Week 12 and Week 24
  Mean change of TSS from baseline.
Pharmacokinetics Parameter (PK): Cmax of INCA035784 | Up to approximately 2 years and 90 days
  Defined as maximum observed plasma concentration of INCA035784.
Pharmacokinetics Parameter: Tmax of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the time to reach the maximum plasma concentration of INCA035784.
Pharmacokinetics Parameter: Cmin of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the minimum observed plasma concentration of INCA035784.
Pharmacokinetics Parameter: AUC(0-t) of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the area under the concentration-time curve up to the last measurable concentration of INCA035784.
Pharmacokinetics Parameter: AUC 0-∞ of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the area under the concentration-time curve from 0 to infinity of INCA035784.
Pharmacokinetics Parameter: CL of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the apparent oral dose clearance of INCA035784.
Pharmacokinetics Parameter: Vz of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the apparent oral dose volume of distribution of INCA035784.
Pharmacokinetics Parameter: t1/2 of INCA035784 | Up to approximately 2 years and 90 days
  Defined as the apparent terminal phase disposition half-life of INCA035784.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (16):
- United States (12):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Stanford University, Palo Alto, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Mayo Clinic-Florida, Jacksonville, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - South Austin Medical Center, Austin, Texas
  - University of Texas Southwestern Medical Center Harold C Simmons Comprehensive Cancer Center Blood, Dallas, Texas
  - Huntsman Cancer Institute At University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Macquarie University Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A study to evaluate INCA035784 in Participants With Myeloproliferative Neoplasms — https://incyteclinicaltrials.com/studies/inca035784-101